CLINICAL TRIAL: NCT03152747
Title: Influence of Posterior Vitreous Detachment on Retinal Detachment After Lens Surgery in Myopic Eyes
Acronym: MYOPRED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Collaborators: ESCRS (Unknown)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principle Investigator, Sponsor, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: Myopred
Record Dates: First submitted 2017-04-19; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Myopia; Cataract; Pseudophakic Retinal Detachment
MeSH Terms: conditions — Myopia; Cataract | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Group A with pre-operative complete posterior vitreous detachment Group A will be invited for one follow-up visit (two months post-operatively) followed up by telephone interviews at one, two, three and five years after surgery to determine occurrence of pseudophakic retinal detachment.
  Examinations: Best corrected Visual Acuity (BCVA) , SD-OCT (spectral domain optical coherence tomography), Ultrasound B-scan (substudy only), Slit lamp examination, telephone interview
  Interventions: Device: ultrasound, b-scan
- B: Group B with no/partial PVD
  Group B will be invited for follow-up examinations at two months, six months and one year after surgery to document occurrence of PVD (if a PVD is present at one of the follow-ups, no more visits are necessary). Two, three and five years after surgery, all patients from group B will be interviewed by telephone, as in group A, to document the occurrence of pseudophakic retinal detachment.
  Examinations: BCVA, SD-OCT, Ultrasound B-scan (substudy only), Slit lamp examination, telephone interview
  Interventions: Device: ultrasound, b-scan

INTERVENTIONS:
Device: ultrasound, b-scan — Some selected centres will participate in a substudy. In the substudy population, if the vitreous cortex is not visible on OCT both in the study eye and the fellow eye, or if the OCT is of poor quality and most likely will not allow definite diagnosis, a B-scan ophthalmic ultrasound will be performed by an experienced examiner. The presence or absence of a PVD in the ultrasound measurement will be recorded in the case report form (CRF). If ultrasonography was not performed, allocation to the groups is based on the staging of the reading centre. Otherwise ultrasonography will be used for final diagnosis and group allocation if the reading centre classifies the OCT as not decisive.

SUMMARY:
Phacoemulsification with implantation of posterior chamber lenses represents the gold standard of care for patients needing lens surgery, but there is an increased risk of developing pseudophakic retinal detachment after surgery. Especially myopic patients have an even higher risk of pseudophakic retinal detachment compared to the general population.

The aim of this multicenter study is to document the presence and/or post-operative development of posterior vitreous detachment (PVD) and to assess its influence on the incidence of retinal detachment (RD) in myopes in a time period of three and five years after lens surgery.

618 eyes of patients scheduled for regular lens surgery will be included, defined by an axial length of 25.0 mm or more. To examine the vitreous status, all patients will receive a comprehensive eye examination pre-operatively, including funduscopy with assessment of a Weiss ring and optical coherence tomography (OCT). Patients will be divided into two groups, group A with pre-operative complete PVD and group B with no/partial PVD. Group A will be invited for one follow-up visit (two months post-operatively) followed up by telephone interviews at one, two, three and five years after surgery to determine occurrence of pseudophakic retinal detachment. Group B will be invited for follow -up examinations at two months, six months and one year after surgery to document occurrence of PVD (if a PVD is present at one of the follow-ups, no more visits are necessary). Two, three and five years after surgery, all patients from group B will be interviewed by telephone, as in group A, to document the occurrence of pseudophakic retinal detachment.

In the recent literature the association between the occurrence of PVD pre-/post-operative and RD after lens surgery is well documented but not described for myopic patients. The results of this multicenter study should help to tackle the problem of RD prediction in myopic patients depending on their pre-operative vitreous status, especially in the setting of refractive lens exchange.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 21 years of age
* Patients scheduled for lens surgery with an axial eye length of 25.0 mm or more
* Availability, willingness, sufficient cognitive awareness to comply with examination procedures
* Ability to sign informed consent

Exclusion Criteria:

* Patients with combined surgery (e.g. combined phacoemulsification and vitrectomy or trabeculectomy or DSAEK)
* Patients with previous intraocular surgery (except any kind of laser surgery e.g. retinopexy, refractive laser surgery)
* Patients with recurrent severe anterior or posterior segment inflammation or uveitis of unknown aetiology, or any disease producing an inflammatory reaction in the eye
* Any ophthalmological pathology with the potential to compromise the measurements (e.g. mature/very dense cataract, fixation difficulties)
* Penetrating ocular trauma
* Previous history of retinal detachment
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Patients participating in another study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: 618. The participants will be selected by the clinical investigators at several ophthalmological centres in Austria, Belgium, Spain, Norway and Sweden. As the study population is already scheduled for cataract surgery / refractive lens exchange, recruitment will be performed directly in these centres at the pre-assessment visits. At this visit, optical biometry is performed and patients with suitable axial eye lengths will be screened. If all inclusion and no exclusion criteria are met the patients will be asked to participate in the trial.
Sampling Method: Probability Sample
Enrollment: 618 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
PVD status | Mid 2023
  Number of patients with preoperative and/or post-operatively developed posterior vitreous detachment (PVD)
Incidence of RD | Mid 2023
  Influence of PVD on the incidence of retinal detachment (RD) in myopes after lens surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria